CLINICAL TRIAL: NCT05513027
Title: A Prospective Study of the Augmented Whole-body Scanning Via Magnifying PET/CT (AWSM-PET/CT) Techniques Abilities to Improve Upon the Diagnostic Accuracy of the Standard-of-care (SOC) PET/CT for Malignant Lesion Detection
Brief Title: Augmented Whole-body Scanning Via Magnifying PET/CT (AWSM-PET/CT) Techniques Abilities to Improve Upon the Diagnostic Accuracy of the Standard-of-care (SOC) PET/CT for Malignant Lesion Detection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202207154; 1R01CA233912 (NIH)
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Magnifying PET; virtual-pinhole PET; cancer; FDG PET/CT
MeSH Terms: conditions — Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Augmented Whole-body Scanning via Magnifying PET (AWSM-PET) (Experimental): All enrolled subjects will undergo SOC PET/CT scan with an AWSM PET device positioned at the far end of the Biograph Vision PET/CT scanner. The patient will receive injection of the PET radiopharmaceutical according to the SOC PET/CT protocol dosing schedule. The entire study will require approximately 2 ½ - 3 hours (from the time patient arrives to the completion of the scan).
  Interventions: Device: Augmented Whole-body Scanning via Magnifying PET; Device: PET/CT

INTERVENTIONS:
Device: Augmented Whole-body Scanning via Magnifying PET — -Added at the end of the SOC PET/CT scan. Will take approximately 3-5 minutes longer.
  Other Names: AWSM-PET
Device: PET/CT — -Standard of care

SUMMARY:
Fluorodeoxyglucose (FDG)-positron emission tomography (PET)/computed tomography (CT) has been demonstrated to outperform other imaging modalities such as CT and magnetic resonance imaging (MRI) for the detection of metastatic cancers. Therefore, it is currently used for cancer staging, re-staging, and for monitoring response to therapy for many types of cancers. Major advances in PET imaging came to the field in 2016, 2020, 2021 and 2023 when the FDA approved additional PET imaging agents to expand the role of cancer detection to include prostate and neuroendocrine cancers. Despite its wide use and success, the diagnostic accuracy of PET/CT is suboptimal for lesions that are significantly smaller than 1 cm due primarily to limitations on image resolution and system sensitivity. The investigators have developed an Augmented Whole-body Scanning via Magnifying PET (AWSM-PET) technology that can improve the image resolution and system sensitivity of current and future PET/CT scanners. This study will evaluate preliminarily whether the AWSM-PET/CT technology can provide additional high-resolution PET/CT images displayed concurrently with the standard of care PET/CT images to improve overall accuracy in depicting malignant lesions in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 years of age or older
* Patient with suspected or pathologically confirmed diagnosis of carcinoma scheduled to undergo standard of care (SOC) PET/CT for initial diagnosis, initial staging, or suspected recurrence. Preference is to enroll those subjects who will undergo biopsy or surgical resection prior to other cancer treatment.
* Willing to undergo PET/CT imaging with AWSM-PET.
* Patients of child-bearing potential must have a negative urine pregnancy test on the day of the PET/CT scan. Postmenopausal women who self-report as amenorrheic for at least 12 consecutive months are to be considered not of child-bearing potential.
* Patients must be able to understand and sign an IRB-approved informed consent form that allows access to prior medical records, participation in the study and chart review follow up.
* Patients are able to tolerate up to approximately 30 min of PET imaging.

Exclusion Criteria:

* For FDG PET/CT only: Patients who have poorly controlled diabetes (fasting blood glucose > 200 mg/dL obtained directly prior to FDG administration for PET/CT scan)
* Patients whose weight or whose body habitus prohibits the AWSM-PET insert device from being placed at the end of the imaging field of view

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
True presence and absence of malignancy in each lesion | Through 9 months after completion of scan
  The true presence and absence of malignancy in each lesion (binary reference standard), will be obtained through multiple sources including pathology report of surgically removed or biopsied tissues, imaging follow-up and clinical follow-up. The separately reconstructed SOC PET/CT and the AWSM PET/CT imaging reading of each lesion will be graded by two raters, separately, via a five-point scale: 1 = definitely benign; 2 = probably benign; 3 = equivocal; 4 = probably malignant; and 5 = definitely malignant. For patients who proceed to surgery or biopsy and histopathologic results are available, the two sets of images with be compared and correlated with the histopathologic results. Each scan will be graded in concordance with the reference standard as true positive, true negative, false positive or false negative. If there is a question about lesion location corresponding to the same area on imaging and pathology additional resources such as the operative report will be utilized.
Image reading of each lesion on SOC PET/CT | Through 45 days after completion of scan
  SOC PET/CT image reading of each lesion, will be graded by two raters, separately, via a five-point scale: 1 = definitely benign; 2 = probably benign; 3 = equivocal; 4 = probably malignant; and 5 = definitely malignant.
Image reading of each lesion on AWSM-PET/CT | Through 45 days after completion of scan
  AWSM PET/CT image reading of each lesion, will be graded by two raters, separately, via a five-point scale: 1 = definitely benign; 2 = probably benign; 3 = equivocal; 4 = probably malignant; and 5 = definitely malignant.

SECONDARY OUTCOMES:
To assess whether a nuclear medicine physician's confidence is altered by the AWSM-PET/CT technology | Through 45 days after completion of scan
  Evaluate whether the indefinite ratings (score of 2-4) for SOC PET/CT is changed to a definitive category (categories 1 and 5) by the AWSM-PET/CT. A study specific review outside of the SOC PET/CT report will be conducted by 2 certified nuclear medicine physicians in batch analyses. The batch analyeses will occur in groups of 3 participants and will be completed within 21 days after the 3rd partcipant's AWSM-PET/CT has been reconstructed. Both physicians will review the SOC PET/CT followed by review of the SOC PET/CT with the AWSM-PET/CT as supplemental imaging. Up to 4 lesions will be recorded and graded according to a five-point scale: 1 = definitely benign; 2 = probably benign; 3 = equivocal; 4 = probably malignant; and 5 = definitely malignant
Image quality score | Through 45 days after completion of scan
  Image quality score of the SOC PET/CT and the AWSM-PET/CT images will be compared to confirm that the simultaneously acquired scans are both of diagnostic quality. A study specific review outside of the SOC PET/CT report will be conducted by 2 certified nuclear medicine physicians in batch analyses. The batch analyeses will occur in groups of 3 participants and will be completed within 21 days after the 3rd partcipant's AWSM-PET/CT has been reconstructed. Both physicians will review the SOC PET/CT followed by review of the SOC PET/CT with the AWSM-PET/CT as supplemental imaging.
  Overall quality of the assigned scan will be evaluated and graded on a 4 point scale: 1= Poor uninterpretable; 2= Poor acceptable for review; 3= Fair; 4= Good/Diagnostic.
Tolerability as measured by number of patients who find the scan intolerable and have to terminate the study | Through completion of study (estimated to be 30 months)
Tolerability as measured by overall comfort of the scan | Through completion of scan (Day 1)
  The overall comfort during the last 3-5 minutes of the scan (added due to the AWSM-PET/CT technology) as compared to the first 15-20 minutes of the scan (for a typical SOC PET/CT). This will be reported via a five-point scale: 1 = extremely uncomfortable, unbearable; 2 = somewhat uncomfortable but bearable; 3 = neutral, neither comfortable nor uncomfortable; 4 = somewhat comfortable; 5 = very comfortable and relaxing.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Chuan Tai, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual patient data that underlie the results reported including text, tables, figures, images and appendices. Study protocol, blank consent, imaging data in DICOM format
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 6 months of initial publication no planned end date
Access Criteria: Anyone who can access the data
URL: https://www.cancerimagingarchive.net/

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu